CLINICAL TRIAL: NCT04254991
Title: A Controlled, Blinded Study to Validate the Diagnostic Accuracy and Assess the Clinical Utility of a Host-response Based Diagnostic Tool for Distinguishing Between Bacterial and Viral Etiologies in Pediatric Patients Presenting to the ED With Suspicion of Acute Infection
Acronym: ROSETTA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MeMed Diagnostics Ltd. (Industry)
Collaborators: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0666-15-RMC
Record Dates: First submitted 2020-01-07; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Viral Infection; Bacterial Infections; Antibiotic Misuse; Host Response Diagnostics
MeSH Terms: conditions — Virus Diseases; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infectious disease group
  Interventions: Diagnostic Test: ImmunoXpert™
- Non-infectious disease group
  Interventions: Diagnostic Test: ImmunoXpert™

INTERVENTIONS:
Diagnostic Test: ImmunoXpert™ — The ImmunoXpert™ technology employs a biochemical assay that measures a proprietary combination of three biomarkers of the immune system coupled with pattern recognition algorithms that classify the source of an infection as bacterial or viral

SUMMARY:
To externally validate the diagnostic accuracy and assess the clinical utility of a host-response based diagnostic tool called ImmunoXpert™, for differentiating between bacterial and viral etiologies in pediatric patients >3 months old with suspicion of Respiratory tract infection (RTI) or Fever without Source (FWS)

ELIGIBILITY:
Inclusion Criteria:

* Documented peak temperature ≥ 38°C (100.4°F) (AND)
* Symptom duration ≤ 7 days (AND)
* Clinical suspicion of RTI (OR)
* Fever without a clear source (OR)
* Acute gastroenteritis (OR)
* Urinary tract infection

Exclusion Criteria:

* Antibiotic treatment of over 48 hours' duration at time of presentation
* Another episode of febrile infection within the past 2 weeks
* A proven or suspected HIV1, HBV, or HCV infection
* Congenital immune deficiency (CID)
* Active malignancy
* Current treatment with immune-suppressive or immune-modulating therapies, including without limitations:

  * Use of high dose steroids >1 mg/kg/day prednisone or equivalent in the past two weeks Monoclonal antibodies, anti-TNF agents
  * Intravenous immunoglobulin (IVIG)
  * Cyclosporine, Cyclophosphamide, Tacrolimus
  * G/GM-CSF, Interferons
* Other severe illnesses that affect life expectancy and quality of life such as:

  * Moderate to severe psychomotor retardation
  * Post-transplant patients
  * Moderate to severe congenital metabolic disorder

Ages: 3 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population will include eligible subjects from both genders that present to the ED due to suspected RTI, FWS, GE, UTI or non-febrile non-infectious disease (Control). Each of these subjects falls into one of the following categories:
  1. Patients with an acute bacterial infection
  2. Patients with an acute viral infection
  3. Patients with an acute mixed co-infection (bacterial and viral)
  4. Patients with an undetermined disease etiology
  5. Patients with a non-infectious disease (control group)
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
ImmunoXpert™ Diagnostic Performance | Through study completion, an average of 3 years
  Sensitivity and specificity of ImmunoXpert™ in differentiating between bacterial and viral etiologies of pediatric patients >3 months old with suspicion of RTI or FWS

SECONDARY OUTCOMES:
ImmunoXpert™ Diagnostic Performance in Pediatric Patients with Gastroenteritis | Through study completion, an average of 3 years
  Sensitivity and specificity of ImmunoXpert in differentiating between bacterial and viral etiologies of pediatric patients >3 months old with GE.
ImmunoXpert™ Diagnostic Performance in Pediatric Patients with Urinary Tract Infection | Through study completion, an average of 3 years
  Sensitivity and specificity of ImmunoXpert in differentiating between bacterial and viral etiologies of pediatric patients >3 months old with UTI.

IPD SHARING:
Plan to Share IPD: No